CLINICAL TRIAL: NCT04471246
Title: High-dose Cephalexin for Cellulitis: A Pilot Randomized Controlled Trial
Brief Title: High-dose vs. Standard-dose Cephalexin for Cellulitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: The Ottawa Hospital Academic Medical Association (Other); Canadian Association of Emergency Physicians (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20200175
Record Dates: First submitted 2020-06-30; First posted 2020-07-15 (Actual); Results first posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-12

CONDITIONS: Cellulitis
MeSH Terms: conditions — Cellulitis | interventions — Cephalexin

STUDY DESIGN:
Intervention Model Description: The Investigators will conduct a parallel arm double-blind randomized controlled pilot trial.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Eligible patients will be randomized (1:1) to high-dose versus standard-dose arms. The randomization sequence will be computer-generated by a statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Dose Cephalexin (Experimental): The intervention is high-dose cephalexin (1000mg PO QID) for seven days
  Interventions: Drug: Cephalexin
- Standard Dose Cephalexin (Active Comparator): The comparator is standard-dose cephalexin (500mg PO QID) plus oral placebo for seven days
  Interventions: Drug: Cephalexin + placebo

INTERVENTIONS:
Drug: Cephalexin — 1000 mg PO QID for 7 days
  Other Names: High-dose cephalexin
  Arms: High Dose Cephalexin
Drug: Cephalexin + placebo — 500 mg PO QID plus oral placebo for 7 days
  Other Names: Standard-dose cephalexin
  Arms: Standard Dose Cephalexin

SUMMARY:
Cellulitis is a painful bacterial infection of the skin and underlying tissue that needs antibiotic treatment. There are approximately 193,000 visits to Canadian emergency departments (EDs) each year for cellulitis. Emergency doctors who treat patients with cellulitis must decide on the correct antibiotic agent, dose, duration and frequency. Cellulitis is most commonly treated with the oral antibiotic cephalexin. However, there has been little research to guide doctors with respect to cellulitis treatment, which has led to an overuse of intravenous antibiotics. In addition, the current treatment failure rate of 20% is unacceptably high. When compared to standard-dose oral cephalexin, high-dose oral cephalexin may reduce treatment failure, which would help decrease the need for intravenous antibiotics and subsequent hospitalization. A well-designed clinical trial is necessary to determine if high-dose oral cephalexin reduces treatment failure for cellulitis patients. This pilot trial will determine the feasibility and design of such a clinical trial.

DETAILED DESCRIPTION:
Background: Cellulitis is a common clinical condition that represents up to 3% of all emergency department (ED) visits. The current treatment failure rate is approximately 20%. This high treatment failure rate may be due to suboptimal dosing of cephalexin. The Investigators hypothesize that high-dose cephalexin may lead to lower rates of treatment failure and subsequently improved patient outcomes (less hospitalizations and avoidance of intravenous antibiotics)

Rationale: Before embarking on a large, multicenter trial, it is essential to conduct a smaller pilot to test and refine study procedures and to demonstrate feasibility.

Methods:

Design: The investigators will conduct a parallel arm double-blind randomized controlled pilot trial at the Civic and General campus ED of The Ottawa Hospital (TOH). The study will operate seven days a week from 0800 to 2000 over a 6-month timeframe. TOH Pharmacy will follow a randomization sequence and prepare study medication packages. Study medication packages will be dispensed to the patient by a registered nurse (RN).

Patients: Adult (age >=18 years) ED patient with non-purulent cellulitis determined by the treating emergency physician to be eligible for outpatient care with oral antibiotics.

Intervention: High-dose cephalexin (1000 mg PO QID) for seven days.

Comparator: Standard-dose cephalexin (500 mg PO QID) plus placebo for seven days.

Primary Feasibility Outcome: Patient recruitment rate (percentage of approached eligible patients who are successfully recruited). The goal is to recruit at least 29% of eligible patients.

Primary Effectiveness Outcome: 1. Oral antibiotic treatment failure, defined as a change in antibiotic (change in class of oral antibiotic or step up to intravenous therapy) within 7 days due to worsening infection, which is defined as:

1. New fever (temperature ≥ 38.0C) or persistent fever at Day 3 follow up; or
2. Increasing area of erythema ≥20% from baseline; or
3. Increasing pain ≥2 points from baseline (numeric rating scale)

The secondary effectiveness outcomes are:

1. Clinical cure (no erythema, pain and fever) at day 7
2. Clinical response (≥20% reduction in area of erythema compared to baseline) at day 3
3. Adverse events (e.g. vomiting, diarrhea, rash) at 14-day telephone follow-up
4. Unplanned i) return ED visits; and ii) hospitalization at 14-day telephone follow-up

Importance: This pilot trial will be the first to compare high-dose cephalexin to standard-dose cephalexin for ED patients with cellulitis. The results of this pilot randomized trial will help inform the design and implementation of a larger, multicenter randomized controlled trial to answer this important clinical question.

ELIGIBILITY:
Inclusion Criteria:

Adults (age >=18 years) with non-purulent cellulitis determined by the treating emergency physician to be eligible for outpatient care with oral antibiotics.

Exclusion Criteria:

1. Age <18 years
2. Patient already taking oral antibiotics
3. Treating physician decides that intravenous therapy is required
4. Abscess requiring an incision and drainage or needle aspiration procedure
5. Known prior cellulitis secondary to methicillin-resistant Staphylococcus aureus
6. Cellulitis secondary to a human or animal bite wound
7. Surgical site infection
8. Malignancy and currently being treated with chemotherapy
9. Febrile neutropenia (temperature >=38C plus absolute neutrophil count <500 cells/uL)
10. Solid organ or bone marrow transplant recipient
11. Renal impairment with creatinine clearance <30 mL/min
12. Pregnant or breastfeeding
13. Allergy to cephalosporins or history of anaphylaxis to penicillin
14. Inability to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2022-02-23 (Actual); Study Completion 2022-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Krishan Yadav, MD, MSc, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stevens DL, Eron LL. In the clinic. Cellulitis and soft-tissue infections. Ann Intern Med. 2009 Jan 6;150(1):ITC11. doi: 10.7326/0003-4819-150-1-200901060-01001. PMID 19124814
- [Result] Stenstrom R, Grafstein E, Romney M, Fahimi J, Harris D, Hunte G, Innes G, Christenson J. Prevalence of and risk factors for methicillin-resistant Staphylococcus aureus skin and soft tissue infection in a Canadian emergency department. CJEM. 2009 Sep;11(5):430-8. doi: 10.1017/s1481803500011623. PMID 19788787
- [Result] Yadav K, Suh KN, Eagles D, MacIsaac J, Ritchie D, Bernick J, Thiruganasambandamoorthy V, Wells G, Stiell IG. Predictors of Oral Antibiotic Treatment Failure for Nonpurulent Skin and Soft Tissue Infections in the Emergency Department. Acad Emerg Med. 2019 Jan;26(1):51-59. doi: 10.1111/acem.13492. Epub 2018 Jul 4. PMID 29869364
- [Result] Pollack CV Jr, Amin A, Ford WT Jr, Finley R, Kaye KS, Nguyen HH, Rybak MJ, Talan D. Acute bacterial skin and skin structure infections (ABSSSI): practice guidelines for management and care transitions in the emergency department and hospital. J Emerg Med. 2015 Apr;48(4):508-19. doi: 10.1016/j.jemermed.2014.12.001. Epub 2015 Jan 17. PMID 25605319
- [Result] Stevens DL, Bisno AL, Chambers HF, Dellinger EP, Goldstein EJ, Gorbach SL, Hirschmann JV, Kaplan SL, Montoya JG, Wade JC; Infectious Diseases Society of America. Practice guidelines for the diagnosis and management of skin and soft tissue infections: 2014 update by the Infectious Diseases Society of America. Clin Infect Dis. 2014 Jul 15;59(2):e10-52. doi: 10.1093/cid/ciu444. PMID 24973422
- [Result] Kwak YG, Choi SH, Kim T, Park SY, Seo SH, Kim MB, Choi SH. Clinical Guidelines for the Antibiotic Treatment for Community-Acquired Skin and Soft Tissue Infection. Infect Chemother. 2017 Dec;49(4):301-325. doi: 10.3947/ic.2017.49.4.301. PMID 29299899
- [Result] Li HK, Agweyu A, English M, Bejon P. An unsupported preference for intravenous antibiotics. PLoS Med. 2015 May 19;12(5):e1001825. doi: 10.1371/journal.pmed.1001825. eCollection 2015 May. PMID 25992781
- [Result] Cyriac JM, James E. Switch over from intravenous to oral therapy: A concise overview. J Pharmacol Pharmacother. 2014 Apr;5(2):83-7. doi: 10.4103/0976-500X.130042. PMID 24799810
- [Result] Yadav K, Gatien M, Corrales-Medina V, Stiell I. Antimicrobial treatment decision for non-purulent skin and soft tissue infections in the emergency department. CJEM. 2017 May;19(3):175-180. doi: 10.1017/cem.2016.347. Epub 2016 Aug 17. PMID 27531595
- [Result] Chow M, Quintiliani R, Cunha BA, Thompson M, Finkelstein E, Nightingale CH. Pharmacokinetics of high-dose oral cephalosporins. J Clin Pharmacol. 1979 Apr;19(4):185-94. doi: 10.1002/j.1552-4604.1979.tb01650.x. No abstract available. PMID 438352
- [Result] Wise R. The pharmacokinetics of the oral cephalosporins--a review. J Antimicrob Chemother. 1990 Dec;26 Suppl E:13-20. doi: 10.1093/jac/26.suppl_e.13. PMID 2292525
- [Result] Murray H, Stiell I, Wells G. Treatment failure in emergency department patients with cellulitis. CJEM. 2005 Jul;7(4):228-34. doi: 10.1017/s1481803500014342. PMID 17355677
- [Result] Peterson D, McLeod S, Woolfrey K, McRae A. Predictors of failure of empiric outpatient antibiotic therapy in emergency department patients with uncomplicated cellulitis. Acad Emerg Med. 2014 May;21(5):526-31. doi: 10.1111/acem.12371. PMID 24842503
- [Result] Yadav K, Nath A, Suh KN, Sikora L, Eagles D. Treatment failure definitions for non-purulent skin and soft tissue infections: a systematic review. Infection. 2020 Feb;48(1):75-83. doi: 10.1007/s15010-019-01347-w. Epub 2019 Aug 5. PMID 31378847
- [Derived] Yadav K, Eagles D, Perry JJ, Taljaard M, Sandino-Gold G, Nemnom MJ, Corrales-Medina V, Suh KN, Stiell IG. High-dose cephalexin for cellulitis: a pilot randomized controlled trial. CJEM. 2023 Jan;25(1):22-30. doi: 10.1007/s43678-022-00433-7. Epub 2023 Jan 2. PMID 36592299

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three randomized patients were excluded due to an alternat diagnosis, thus 66 moved forward for analysis (33 in each arm)
Groups:
- Standard Dose Cephalexin: The comparator is standard-dose cephalexin (500mg PO QID) plus oral placebo for seven days
  Cephalexin: 500 mg PO QID plus oral placebo for 7 days
Period: Overall Study
Arm/Group | High Dose Cephalexin | Standard Dose Cephalexin
Started | 33 | 33
Completed | 31 | 31
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose Cephalexin | Standard Dose Cephalexin | Total
Number analyzed (Participants) | 33 | 33 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 2
  Between 18 and 65 years | 19 | 22 | 41
  >=65 years | 13 | 10 | 23
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 56 [34 to 71] | 57 [40 to 69] | 56 [37 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 20 | 20 | 40
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 33 | 33 | 66
BMI [Median (Inter-Quartile Range); unit: kg/m2] | 30.4 [24.4 to 36.8] | 27.9 [23.4 to 31.6] | 29.1 [24.1 to 34.6]
Height [Median (Inter-Quartile Range); unit: metres] | 1.72 [1.63 to 1.8] | 1.67 [1.59 to 1.79] | 1.7 [1.62 to 1.8]
Weight [Median (Inter-Quartile Range); unit: kg] | 90 [76.5 to 106.5] | 80 [64 to 96.5] | 84.5 [74 to 100]

OUTCOME MEASURES:

1. Primary Outcome: Patient Recruitment Rate
Description: % of patients recruited into the trial
Time Frame: 6 months
Population: Number of patients within the 6 months of the trial that were determined to be eligible of the trial. Of 134, 69 were successfully approached and recruited in the study.
Measure: Number; unit: percentage of eligible patients
Groups:
- Patients Identified as Eligible for the Trial: Total number of participants deemed eligible for the study
Arm/Group | Patients Identified as Eligible for the Trial
Number analyzed (Participants) | 134
percentage of eligible patients | 51.5

2. Primary Outcome: Oral Antibiotic Treatment Failure
Description: % of patients with oral antibiotic treatment failure
  Oral antibiotic treatment failure, defined as a change in antibiotic (change in class of oral antibiotic or step up to intravenous therapy) within 7 days due to worsening infection, which is defined as:
  1. New fever (temperature ≥ 38.0°C) or persistent fever at Day 3 follow up; or
  2. Increasing area of erythema ≥20% from baseline; or
  3. Increasing pain ≥2 points from baseline (numeric rating scale)
Time Frame: Each patient was assessed for oral antibiotic treatment failure at the day 3 and day 7 follow-ups
Population: Of 66 patients enrolled and confirmed to have cellulitis by the Principal Investigator, 62 were assessed for treatment failure. Four were lost to follow-up and therefore could not be assessed for treatment failure.
Measure: Number (95% Confidence Interval); unit: percentage of enrolled in each arm
Arm/Group | High Dose Cephalexin | Standard Dose Cephalexin
Number analyzed (Participants) | 31 | 31
percentage of enrolled in each arm | 3.2 [0.6 to 16.2] | 12.9 [5.1 to 28.9]

3. Secondary Outcome: Ability to Approach Eligible Patients
Description: % of eligible patients that were identified as being eligible but missed (staff was unable to approach to recruit in trial)
Time Frame: 6 months
Measure: Number; unit: percentage of eligible patients
Groups:
- Patients Identified as Eligible for the Trial: Participants that after screening were determined to be eligible for the trial
Arm/Group | Patients Identified as Eligible for the Trial
Number analyzed (Participants) | 134
percentage of eligible patients | 14.2

4. Secondary Outcome: Assessment of Blinding
Description: The percentage of patients that correctly guessed their treatment allocation.
  To assess how well blinded the patients were to the medication they received, each was asked during the day 7 follow-up, after having finished their medication, to indicate which treatment they believe they received (500mg of 1000mg of cephalexin). Once unblinded to the allocation (after enrollment and follow-up complete), it was possible to determine which patients correctly guess the dose of medication they received.
Time Frame: Patient were asked which dose of cephalexin they believe they received during the day 7 follow-up
Measure: Number; unit: percentage of enrolled per arm
Groups:
- High-dose Group: Patient enrolled in the trial with a confirmed diagnosis of cellulitis that received high-dose cephalexin (1000mg PO four times a day for 7 days)
- Standard-dose Group: Patient enrolled in the trial with a confirmed diagnosis of cellulitis that received standard-dose cephalexin (500mg + placebo) PO four times a day for 7 days)
Arm/Group | High-dose Group | Standard-dose Group
Number analyzed (Participants) | 33 | 33
percentage of enrolled per arm | 33.3 | 60.1

5. Secondary Outcome: Protocol Adherence
Description: % of patients that are adherent to allocated treatment for 7 days
Time Frame: 7 days
Measure: Number; unit: percentage of enrolled and analyzed
Groups:
- Standard-dose Group: Patient enrolled in the trial with a confirmed diagnosis of cellulitis that received standard-dose cephalexin (500mg + placebo PO four times a day for 7 days)
Arm/Group | High-dose Group | Standard-dose Group
Number analyzed (Participants) | 33 | 33
percentage of enrolled and analyzed | 75.8 | 75.8

6. Secondary Outcome: Loss to Follow-up
Description: % of patients lost to follow-up at 14 days
  Patients were lost to follow-up if they did not attend any follow-up visit at days 3, 7 and 14
Time Frame: Determined at final follow-up (day 14) if lost to follow-up
Measure: Number; unit: percentage of enrolled per arm
Arm/Group | High-dose Group | Standard-dose Group
Number analyzed (Participants) | 33 | 33
percentage of enrolled per arm | 6.1 | 6.1

7. Secondary Outcome: Clinical Cure
Description: % of patients with clinical cure (no erythema, pain and fever) at days 7 and 14
Time Frame: Assessed for clinical cure at day 7and day 14 follow-up
Population: Of the 66 enrolled and confirmed to have cellulitis, 4 were lost to follow-up. The remaining 62 were analyzed for clinical cure at days 7 and 14.
Measure: Number (95% Confidence Interval); unit: percentage of enrolled in each arm
Arm/Group | High Dose Cephalexin | Standard Dose Cephalexin
Number analyzed (Participants) | 31 | 31
percentage of enrolled in each arm
  Clinical cure at day 14 | 45.2 [29.2 to 62.2] | 38.7 [23.7 to 56.2]
  Clinical cure at day 7 | 16.1 [7.1 to 32.6] | 6.5 [1.8 to 20.7]

8. Secondary Outcome: Adverse Events
Description: % of patients with adverse events (e.g. vomiting, diarrhea, rash) at 14-days measured via telephone follow-up
Time Frame: 14 days
Population: Of the 66 enrolled and confirmed to have cellulitis, 4 were lost to follow-up. The remaining 62 were assessed for adverse events.
Measure: Number (95% Confidence Interval); unit: percentage of enrolled in each arm
Arm/Group | High Dose Cephalexin | Standard Dose Cephalexin
Number analyzed (Participants) | 31 | 31
percentage of enrolled in each arm
  Nausea or vomiting | 9.7 [3.4 to 24.9] | 3.2 [0.6 to 16.2]
  Diarrhea | 16.1 [7.1 to 32.6] | 6.5 [1.8 to 20.7]
  Abdominal pain | 3.2 [0.6 to 16.2] | 0 [0 to 11]
  Rash | 3.2 [0.6 to 16.2] | 6.5 [1.8 to 20.7]
  Other | 6.5 [1.8 to 20.7] | 9.7 [3.4 to 24.9]
  No adverse events to report | 61.3 [43.8 to 76.3] | 74.2 [56.8 to 86.3]

9. Secondary Outcome: Unplanned ED Visits or Hospitalization
Description: % of patients with unplanned i) return ED visits; and ii) hospitalization, measured via 14-day telephone follow-up
Time Frame: 14 days
Population: Of the 66 enrolled and confirmed to have cellulitis, 4 were lost to follow-up. The remaining 62 were assessed for unplanned ED visit or hospitalizations at the day 14 telephone follow-up
Measure: Number (95% Confidence Interval); unit: percentage of enrolled in each arm
Arm/Group | High Dose Cephalexin | Standard Dose Cephalexin
Number analyzed (Participants) | 31 | 31
percentage of enrolled in each arm
  Unplanned visit to family doctor within 14 days | 6.5 [1.8 to 20.7] | 6.5 [1.8 to 20.7]
  Unplanned return to ED within 14 days | 22.6 [11.4 to 39.8] | 16.1 [7.1 to 32.6]
  Unplanned hospitalization within 14 days | 0 [0 to 11] | 0 [0 to 11]

ADVERSE EVENTS:
Time Frame: Patients were assessed for adverse events during the day 7 and day 14 study follow-ups
Arm/Group | High Dose Cephalexin | Standard Dose Cephalexin
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 12/31 | 8/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High Dose Cephalexin (N=31) | Standard Dose Cephalexin (N=31)
Nausea or vomiting (Gastrointestinal disorders) | 3 | 1
Diarrhea (Gastrointestinal disorders) | 5 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 — Rash that has developed after starting the medication
Other (Product Issues) | 2 | 3 — Any other non-serious adverse event reported by patient that was not included in the list of adverse events captured in the patient questionnaires

LIMITATIONS AND CAVEATS:
A small proportion of participants who reported clinical cure at the end-of-therapy visit. We have recently published a systematic review that demonstrates that symptoms such as pain and erythema can persist beyond 14 days.

We were unable to assess for infection recurrence beyond 14 days. We will mitigate this in a future trial by including a 30-day telephone follow-up.

Secondary feasibility target of < 10% missed eligible patients not met.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-24): https://cdn.clinicaltrials.gov/large-docs/46/NCT04471246/Prot_SAP_000.pdf